CLINICAL TRIAL: NCT05586958
Title: A Randomized, Multi-regional, Double-blind, Parallel-group, Placebo-controlled Phase 3 Study to Assess the Safety and Efficacy of 6 Months Treatment With Tigulixostat in Gout Patients With Hyperuricemia
Brief Title: Tigulixostat, Phase 3 Study, Placebo Controlled in Gout Patients
Acronym: EURELIA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-GDCL009
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Gout; Hyperuricemia; Gout Flare; Tophi
Keywords: Gout; Hyperuricemia; Xanthine Oxidase Inhibitor
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tigulixostat 100mg (Experimental): Tigulixostat 100mg, Once a day (QD) for up to 6 months
  Interventions: Drug: Tigulixostat
- Tigulixostat 200mg (Experimental): Tigulixostat 200mg, Once a day (QD) for up to 6 months
  Interventions: Drug: Tigulixostat
- Tigulixostat 300mg (Experimental): Tigulixostat 300mg (100mg + 200mg), Once a day (QD) for up to 6 months
  Interventions: Drug: Tigulixostat
- Placebo (Placebo Comparator): Placebo, Once a day (QD) for up to 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tigulixostat — Xanthine Oxidase Inhibitor
  Other Names: LC350189
  Arms: Tigulixostat 100mg; Tigulixostat 200mg; Tigulixostat 300mg
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The aim of this 6-month randomized multi-regional double-blind parallel group placebo-controlled phase 3 study is to assess the efficacy and safety of three different doses of Tigulixostat in gout patients with hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 85 years, inclusive.
* Subjects with hyperuricemia and a history or presence of gout per American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2015 criteria.
* Subjects who are currently on urate-lowering therapies (ULT) with an sUA level ≥6.0 mg/dL at screening (Visit 1); or subjects who are currently not on ULT with an sUA level ≥7.0 mg/dL at screening (Visit 1). Subjects currently on ULT will undergo washout and must have an sUA level ≥7.0 mg/dL at Visit 3 to be randomized and participate in the study.
* Subjects with a Body Mass Index ≤50 kg/m2 and estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 at screening (Visit 1).

Exclusion Criteria:

* Subjects with secondary hyperuricemia, enzymatic defects.
* Subjects experiencing an acute gout attack (intense pain, swelling, or/and tenderness in the joint area) within 2 weeks prior to screening (Visit 1).
* Subjects who have received pegloticase to treat gout which has not responded to the usual treatments.
* Subjects who have not been receiving stable doses of drugs known to affect sUA levels for the last 3 weeks prior to screening (Visit 1).
* Subjects with a history of xanthinuria (elevated levels of xanthine in the urine) and rheumatoid arthritis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with sUA levels <6.0 mg/dL sustained at months 4, 5, and 6 | Up to Month 6
  Serum uric acid (sUA) level will be measured at Month 4,5, and 6

SECONDARY OUTCOMES:
The proportion of subjects with sUA levels <5.0 mg/dL sustained at months 4, 5, and 6 | Up to Month 6
  Serum uric acid (sUA) level will be measured at Month 4,5, and 6
The proportion of subjects reporting a gout flare up to each visit. | Up to Month 6
  Gout flare (intense pain, swelling, or/and tenderness in the joint area) will be assessed from baseline up to 6 months
Incidence rate of adverse event | Up to Month 6
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Hyungjin Cho, MD, Study Director — LG Chem
Locations (52):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Medvin Clinical Research, Covina, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Herco Medical and Research Center, Inc, Coral Gables, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Vista Clinical Research, LLC, Newnan, Georgia
  - Velocity Clinical Research, Meridian, Idaho
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - MD Medical Research, Oxon Hill, Maryland
  - Elite Clinical Research, LLC, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Practice Dr. David Headley, Port Gibson, Mississippi
  - HealthCare Research, Hazelwood, Missouri
  - Healor Primary Care/CCT Research, Las Vegas, Nevada
  - Meridian Clinical Research, LLC, Vestal, New York
  - Triad Clinical Trials, Greensboro, North Carolina
  - STAT Research, Vandalia, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Tristar Clinical Investigations, P.C., Philadelphia, Pennsylvania
  - Velocity Clinical Research Greenville, Greenville, South Carolina
  - PCCR Solutions, Colleyville, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - South Ogden Family Medicine/CCT Research, South Ogden, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Meridian Clinical Research, LLC, Portsmouth, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
- Georgia (6):
  - LTD "Clinic LJ", Kutaisi
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - LTD Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
  - JSC "Vian", Tbilisi
  - LTD MediClub Georgia, Tbilisi
  - LTD Multiprofile Clinic Consilium Medulla, Tbilisi
- Philippines (6):
  - Angeles University Foundation Medical Center, Angeles
  - Davao Doctors Hospital, Davao City
  - Lipa Medix Medical Center, Lipa
  - Makati Medical Center, Makati
  - Manila Doctors Hospital, Manila
  - ManilaMed - Medical Center, Manila
- Thailand (4):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Bangkoknoi
  - Thammasat University Hospital, Khlong Luang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saag KG, Dalbeth N, Hsu CY, Kuo CF, Nuki G, Perez-Ruiz F, White WB, Hariri A, Lee Y, Jang Y, Han S, Choi HK. Evaluation of the efficacy and safety of a novel xanthine oxidase inhibitor, tigulixostat, in gout patients with hyperuricemia: Design of the EURELIA 1 and EURELIA 2 studies. Contemp Clin Trials. 2025 Apr;151:107843. doi: 10.1016/j.cct.2025.107843. Epub 2025 Feb 8. PMID 39929260